CLINICAL TRIAL: NCT00895518
Title: Effects of Early Psychological Intervention to Prevent PTSD
Brief Title: Examining the Effectiveness of an Early Psychological Intervention to Prevent Post-Traumatic Stress Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Barbara O. Rothbaum, PhD, Professor in Psychiatry and Associate Vice Chair of Clinical Research, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00009260; DATR AD-TS (Other: Other); R34MH083078 (NIH)
Record Dates: First submitted 2009-05-07; First posted 2009-05-08 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (No Intervention): Participants will receive assessments only.
- 2 (Experimental): Participants will receive prolonged exposure therapy.
  Interventions: Behavioral: Prolonged Exposure (PE) Therapy

INTERVENTIONS:
Behavioral: Prolonged Exposure (PE) Therapy — Three PE sessions lasting 1 hour each, delivered 1 week apart
  Arms: 2

SUMMARY:
This study will examine the use of prolonged exposure therapy on people who have recently experienced a trauma to prevent them from developing post-traumatic stress disorder.

DETAILED DESCRIPTION:
Post-traumatic stress disorder (PTSD) is a disorder that forms in response to a traumatic event. The symptoms of PTSD, such as hyper-arousal and re-experiencing the traumatic event, are common in all people who have recently experienced a trauma, but those who develop PTSD continue to have these symptoms more than a month after the trauma. Some researchers believe that developing PTSD is the result of a failure to adequately recover from the trauma. This study will determine whether providing a common form of treatment for PTSD, prolonged exposure (PE) therapy, to people who have recently experienced trauma will prevent them from developing PTSD. The study will also seek to identify predictive markers, such as hormone levels and genes, for developing PTSD.

Participation in this study will last 3 months. Participants will first undergo an evaluation session that will include an interview, questionnaires, and a medical chart review for blood pressure and heart rate measurements taken after their trauma. They will then be randomly assigned to receive either PE therapy or assessments only. Participants receiving PE therapy will complete three weekly treatment sessions, with the first occurring immediately after the evaluation session. Treatment will involve reviewing memories of a recent trauma out loud with a therapist and audio-recording these discussions for review at home. All participants will undergo assessments 1 and 3 months after the initial evaluation session. The 1-month assessment will involve an interview and questionnaires similar to the evaluation session, and the 3-month session will involve only a brief phone interview. Some participants will also be asked to complete an optional part of the study in which they provide two saliva samples to researchers: one to measure stress hormones and one to test for genetic bases of trauma response.

ELIGIBILITY:
Inclusion Criteria:

* Presenting to the emergency department of Emory University School of Medicine/Grady Memorial Hospital for rape in the past 72 hours
* Meets DSM-IV diagnostic criterion A in which both of the following are present: (i) The person experienced, witnessed, or was confronted with an event or events that involved actual or threatened death or serious injury or a threat to the physical integrity of self or others (ii) The person's response involved intense fear, helplessness, or horror
* Speaks and understands spoken English
* Can see the assessment forms, hear instructions, and function at an emotional and intellectual level sufficient to allow accurate completion of all assessment instruments
* No significant traumatic injuries, as determined by the physician

Exclusion Criteria:

* Current or history of mania, schizophrenia, or other psychoses
* Current (past month) prominent suicidal ideation or recent (past 3 months) parasuicidal behavior or other self-injurious behavior, such as low lethality cutting
* Current (past month) substance dependence; people who meet criteria for current substance abuse but not dependence, or past dependence and have been in remission for at least 1 month are eligible.
* Experienced a loss of consciousness for more than 5 minutes as a result of injuries sustained during the trauma
* Intoxicated, altered, or highly distressed to the degree that accurate completion of the study assessments or participation in study procedures is not possible
* Blood alcohol level above .08, determined by breathalyzer in the emergency department
* Not alert, oriented, and coherent
* In severe pain, active labor, or respiratory distress or hemodynamically compromised in any way

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2008-04; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
PTSD Symptom Scale- I (PSS) | Measured 4 and 12 weeks post-trauma

CONTACTS AND LOCATIONS:
Overall Officials: Barbara O. Rothbaum, PhD, Principal Investigator — Emory University
Locations (1):
- Grady Memorial Hospital, Emergency Department, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Rothbaum BO, Kearns MC, Reiser E, Davis JS, Kerley KA, Rothbaum AO, Mercer KB, Price M, Houry D, Ressler KJ. Early intervention following trauma may mitigate genetic risk for PTSD in civilians: a pilot prospective emergency department study. J Clin Psychiatry. 2014 Dec;75(12):1380-7. doi: 10.4088/JCP.13m08715. PMID 25188543
- [Derived] Price M, Kearns M, Houry D, Rothbaum BO. Emergency department predictors of posttraumatic stress reduction for trauma-exposed individuals with and without an early intervention. J Consult Clin Psychol. 2014 Apr;82(2):336-41. doi: 10.1037/a0035537. Epub 2014 Feb 3. PMID 24491070
- [Derived] Rothbaum BO, Kearns MC, Price M, Malcoun E, Davis M, Ressler KJ, Lang D, Houry D. Early intervention may prevent the development of posttraumatic stress disorder: a randomized pilot civilian study with modified prolonged exposure. Biol Psychiatry. 2012 Dec 1;72(11):957-63. doi: 10.1016/j.biopsych.2012.06.002. Epub 2012 Jul 4. PMID 22766415